CLINICAL TRIAL: NCT04616794
Title: Tailored, Multidomain, and Coach-assisted Interactive Mobile Application for the Adoption and Maintenance of a Healthy Lifestyle in Middle-aged and Older Adults With Modifiable Risk Factors for Dementia: A Proof-of-concept Study
Brief Title: Intervention on Modifiable Lifestyle Risk Factors for Dementia Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LuciLab (Industry)
Collaborators: Centre de Recherche de l'Institut Universitaire de Geriatrie de Montreal (Other); Sojecci II Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LUCI-01
Record Dates: First submitted 2020-10-13; First posted 2020-11-05 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2021-02

CONDITIONS: Risk Behavior; Cognitive Decline
MeSH Terms: conditions — Risk-Taking; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: The Luci intervention is a personalized lifestyle behaviour change program delivered via an interactive mobile platform with the online support of a coach. The system will allow participants to communicate with their coach through video calls and a messaging/chat system. The coaching sessions will focus on providing personalized support to help participants improve their eating habits, cognitive engagement and/or physical activity. The coach will offer assistance, feedback, information where appropriate, and motivational support throughout the trial. The Proof-of-Concept study is a 10-week pre-post within-subject parallel group treatment-only study. There will be three single-domain groups, and one multidomain group. Participants will receive coach-assisted counselling for up to 9 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cognitive Engagement Group (Experimental): Participants eligible to enter this group must show low cognitive engagement in cognitively stimulating activities, defined as a score < 22 on the Cognitive Activity Questionnaire (CAQ)
  Interventions: Behavioral: Cognitive Engagement Group
- Physical Activity Group (Experimental): Participants eligible to enter this group must have a low level of physical activity defined as less than 600 MET-min/week (~150 minutes/week) of moderate to vigorous physical activity (MVPA), measured using the International Physical Activity Questionnaire - short form (IPAQ-SF)
  Interventions: Behavioral: Physical Activity Group
- Diet Group (Experimental): Participants eligible to enter this group must have a low adherence to the Mediterranean-type diet defined as a score of ≤ 8 on the adapted Canadian Mediterranean Diet Scale (MDS).
  Interventions: Behavioral: Diet Group
- Multi-modal Group (Experimental): Participants eligible to enter this group must be eligible for at least two of the three single-arm conditions.
  Interventions: Behavioral: Multimodal group

INTERVENTIONS:
Behavioral: Cognitive Engagement Group — Participants in this group will be encouraged to lead a cognitively stimulating lifestyle, as a means for cognitive decline/dementia risk reduction. This will be achieved by providing educational materials, practical tips and strategies, and suggestions about the different options to increase cognitively stimulating activities and by assisting participants outlining goals to progressively adopt a more cognitively active lifestyle.
  Arms: Cognitive Engagement Group
Behavioral: Physical Activity Group — Participants in this group will be encouraged to lead a physically active lifestyle, as a means for cognitive decline/dementia risk reduction. This will be achieved by providing educational materials, practical tips and strategies, and suggestions about the different options to increase physical activities and by assisting participants outlining goals to progressively adopt a more physically active lifestyle.
  Arms: Physical Activity Group
Behavioral: Diet Group — Participants in this group will be encouraged to adopt a healthy diet, as a means for cognitive decline/dementia risk reduction. This will be achieved by providing educational materials, practical tips and strategies, and suggestions about the different options to change their diet and by assisting participants outlining goals to progressively adopt a Mediterranean-like diet.
  Arms: Diet Group
Behavioral: Multimodal group — Participants assigned to this group will select which domain they wish to tackle first. Interventions are as described for the single-domain interventions.
  Arms: Multi-modal Group

SUMMARY:
The overarching aim is to develop and deploy a multidomain intervention delivered on a mobile application to help older adults reduce their risk for dementia by improving a set of modifiable lifestyle risk factors associated with cognitive decline/dementia. The targeted domains are physical activity, diet, and cognitively stimulating activity. This registration concerns the Proof-of-concept study which will examine if individual parts of the intervention program achieve a clinically significant degree of change in the targeted behavioral risk outcomes. It is expected that following the program, at least 50% of participants will show evidence of a clinically significant degree of change in the behavioral risk outcome targeted by the intervention, when compared to baseline.

DETAILED DESCRIPTION:
There are encouraging indications from observational and prospective studies that late life multidomain lifestyle interventions can reduce the risk of cognitive decline and dementia, as well as improve cognition. However, these studies raise major issues related to scalability and adherence which can be addressed by relying on technology. These studies mainly used intensive and costly face-to-face interventions that are not easily implemented on a large scale. Furthermore, there are challenges with the adherence to all the components of a multi-domain lifestyle program.

Technology-delivered interventions have the potential to overcome some of the limitations of traditional face-to-face interventions. They confer numerous advantages including scalability of use in a real-world setting while limiting geographical constraints and other logistical challenges such as clinic attendance requirements. Such delivery modes also offer user convenience (e.g., undertaken at home and flexible schedule) and reduced costs associated with large-scale deployment of studies and programs.

In addition to the inclusion of technology, the success of health promotion interventions may also be improved by integrating models of lifestyle habit patterns and behaviour change determinants. The coach-based intervention will integrate behavioural change techniques based on the Behaviour Change Wheel developed by Michie. The coach intervention approach will also be guided by the Transtheoretical model of behaviour change principles proposed by Prochaska and DiClemente, and Motivational Interviewing techniques described by Rollnick and Miller.

The Proof-of-Concept study is a 10-week pre-post within-subject parallel group treatment-only study. There will be three single-domain groups (diet; physical activity or cognitive engagement), and one multidomain group. Participants will receive up to 9 weekly coach-assisted counselling sessions. The goal is to recruit up to 55 participants with at least one of the target risk factors : unhealthy diet, low level of cognitively stimulating activity or physical activity). Participants with a single risk factor will be invited to the single-domain condition for which they have a risk. Participants with multiple risk factors will be invited to the multidomain condition. The risk level for each domain will be examined before and after the intervention to assess whether the intervention has induced a clinically significant change.

ELIGIBILITY:
Inclusion Criteria:

* Proficient or native speakers in French;
* Computer literate;
* Committed not to participate in another program related to any of the three intervention domains for the duration of the trial;
* At least one of the following:

  * Low cognitive engagement in cognitively stimulating activities, defined as a score ≤ 15 on the CAQ
  * Low level of physical activity defined as less than 600 MET-min/week (~150 minutes/week) of MVPA measured using the IPAQ-SF
  * Low adherence to the Mediterranean-type diet defined as a score of ≤ 8 on the adapted Canadian MDS

Exclusion Criteria

* Presence of a cognitive impairment as measured by the Cogstate Brief BatteryTM ;
* General anesthesia within the last 6 months;
* Participation in any previous validation studies related to the program;
* Participation, currently or within the last 6 months, in a program where they received any of the three interventions;
* Unable to commit participation over the period of the study.
* Participants in the precontemplation stage of change.
* Participants with a high level of perceived stress.
* Having received a diagnosis of:

  * Dementia or neurodegenerative disease;
  * Past or present neurological disorder;
  * Severe psychiatric disorder;
  * Uncontrolled cardiovascular or metabolic diseases;
  * Alcoholism or drug addiction;
  * Any other conditions expected to limit participation.

Domain-Specific exclusion criteria

* Participants will be excluded from the physical activity intervention, but not the trial, if they have a medical contraindication to physical activity based on the Physical Activity Readiness Questionnaire
* Individuals with dietary restrictions due to medical reasons, allergies or severe intolerance or an history of eating disorders will be excluded from participation in the healthy diet intervention.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2020-10-13 (Actual); Primary Completion 2020-12-24 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Cognitive Engagement at study end | Baseline (within 1 week before the first coaching session) and study end (within 1 week after the last coaching session)
  Cognitive engagement is measured using the Cognitive Activity Questionnaire (CAQ). Participants are asked to indicate the frequency in which they engage in 10 cognitive leisure activities. Scores range from 0 to 70. A higher score represents a higher cognitive engagement level.
Change from Baseline in Mediterranean Diet Adherence at study end | Baseline (within 1 week before the first coaching session) and study end (within 1 week after the last coaching session)
  Adherence to the Mediterranean Diet is measured with an adaptation of the Canadian Mediterranean Diet Scale (MDS). The scale consists of 13 questions on food consumption frequency and intake habits. Scores range from 0 to 13, where a higher score represents a higher adherence level.
Change from Baseline in Physical Activity at study end | Baseline (within 1 week before the first coaching session) and study end (within 1 week after the last coaching session)
  Physical activity level is measured using the International Physical Activity Questionnaire - Short Form (IPAQ-SF). The IPAQ-SF consists of 7 items to assess Moderate to vigorous physical activity (MVPA) as well as walking and sitting time in the last 7 days. An overall total physical activity score is computed in Metabolic equivalent tasks (MET)-minutes/week, where a higher MET value represents a higher level of physical activity.

SECONDARY OUTCOMES:
Change from Baseline in Luci Cognitive Engagement Score at study end | Baseline (within 1 week before the first coaching session) and study end (within 1 week after the last coaching session)
  Six questions are added to the Cognitive Activity Questionnaire to include stimulating cognitive activities not covered in the original questionnaire. From the whole questionnaire, a total score is computed ranging from 0 to 112, where a higher score represents a higher cognitive engagement level.
Change from Baseline in Luci Mediterranean Diet Adherence Score at study end | Baseline (within 1 week before the first coaching session) and study end (within 1 week after the last coaching session)
  Eight questions are added to the Canadian Mediterranean Diet questionnaire to include food groups and food intake habits not covered in the original questionnaire. From the whole questionnaire, a total score is computed ranging from 0 to 36, where a higher score represents a higher adherence level.
Change from Baseline in Luci Physical Activity Score at study end | Baseline (within 1 week before the first coaching session) and study end (within 1 week after the last coaching session)
  Three questions assess frequency and intensity of specific physical activities related to aerobic, resistance and flexibility training over the past 7 days. Three subscores and a total score ranging from 0-30 are computed, where higher scores represent higher physical activity levels.
Goal Attainment | Weekly (within 1 week after the first coaching session) up to study end (within 1 week after the last coaching session)
  For each goal, level of attainment and perceived effort towards goal attainment are rated weekly using a 10-point Likert-like scale, where 10 represents "completed" and "maximal effort", respectively.
Perceived Progress in adopting lifestyle changes | Study end (within 1 week after the last coaching session)
  Perceived Progress in adopting lifestyle changes will be investigated with a single question, "To what extent do you think you changed your (domain specified) lifestyle since the beginning of the program?", using a 10-point Likert-like scale, where 10 represents a major change.
Change from Baseline in Readiness to change at study end | Baseline (within 1 week before the first coaching session) and study end (within 1 week after the last coaching session)
  Readiness to change will be determined using a 6-item questionnaire at Baseline and a 3-item questionnaire at study end.
Program Quality | Study end (within 1 week after the last coaching session)
  The quality of the program is assessed using the end-user version of the Mobile App Rating Scale (uMARS). The uMARS is a 20-item questionnaire that includes 4 objective quality subscales (engagement, functionality, aesthetics, and information quality), and 1 subjective quality subscale. A summary score is calculated as the mean score across the 4 objective criteria. One further subscale, consisting of 6 items, measures users' perceived impact of the evaluated app. Score range from 0-5, where 5 represents a higher quality and impact, respectively.
Program Usability | Study end (± 1 week after the last coaching session)
  The usability of the program is assessed using the System Usability Scale (SUS). The SUS is a 10-item questionnaire. Scores range from 0-5, where a higher score represents a higher usability.
Satisfaction and Continuance Usage Intention | Study end (within 1 week after the last coaching session)
  The user's continuance intention is assessed using the Satisfaction and Continuance Usage Intention Questionnaire. The questionnaire comprises 28 questions assessing 9 constructs, (Continuance intention, Expectation confirmation, Satisfaction, Perceived usefulness, Perceived ease of use, Trust/Credibility, Perceived security and confidentiality, Perceived service quality, Perceived system quality). Score range from 0-5, where a higher score represent a higher agreement, respectively.
Overall User Experience | Study end (within 1 week after the last coaching session)
  Feedback about the overall user experience with the platform will be collected using a semi-structured interview conducted by phone.
Platform usage | Baseline (within 1 week before the first coaching session) to study end (within 1 week after the last coaching session)
  Continuous measures of different parameters linked to platform usage during the study period will be recorded and analyzed, including pattern of use (e.g., time of day), frequency (e.g., number of platform access), duration of use (e.g., duration of the coach sessions) and the functionalities used (e.g., content viewed).

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie Belleville, PhD, Principal Investigator — Centre de recherche de l'Institut Universitaire de gériatrie de Montréal
Locations (1):
- Sylvie Belleville, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No